CLINICAL TRIAL: NCT03909347
Title: PLAN: Dementia Literacy Education and Navigation for Korean Elders With Probable Dementia and Their Caregivers
Acronym: PLAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); NYU Langone Health (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB00242241; R01AG062649-01 (NIH)
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Dementia
Keywords: Korean American elders; Caregivers; dementia Literacy education And Navigation; Community health workers; successful aging; PLAN
MeSH Terms: conditions — Dementia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Our study will use PRECEDE-PROCEED model for planning and evaluation of interventions to address our intervention delivery model using trained community health workers (CHWs) and community-participatory approaches. Predisposing factors of sociodemographic characteristics like caregiver age, gender, level of education, and English proficiency and the KA elder's Clinical Dementia Rating (CDR) score will be considered as covariates. Enabling factors for the study include caregiver's dementia literacy and self-efficacy in dementia care, and the KA elder's access to medical care, and reinforcing factors include social support and primary physician recommendation for cognitive testing.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLAN (intervention) (Experimental): Group 1 will receive the study intervention during the 6 months of the study, after the first baseline questionnaire. The intervention is as follows: participants will be asked to take part in a one-time, one-hour education in participants' home or any community location that is most convenient for the participants by a trained community health worker. An educational resource that participants can read at home will be provided at the end of education session. Participants' community health worker will call the participants monthly to identify barriers to dementia care and help participants and participants' elder with making an appointment or transportation to the health care facility, when participants request for assistance.
  Interventions: Behavioral: PLAN
- Standard of care (control) (Active Comparator): Group 2 will receive a signs and treatment of dementia pamphlet by the Alzheimer's Association and will be referred to the elder's primary physician.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: PLAN — The study intervention, PLAN is a multifaceted intervention led by trained CHW. It consists of two main components: dementia literacy education and phone counseling with navigation assistance through (1) 1-hour visit for dementia literacy education and (2)monthly counseling with navigation assistance
  Arms: PLAN (intervention)
Behavioral: Standard of Care — The investigators will refer control group participants to participants' primary physicians for follow-up and provide an Alzheimer's Association brochure about signs of dementia and dementia treatment, which is publicly available in Korean.
  Arms: Standard of care (control)

SUMMARY:
Studies have shown that ethnic-racial minority elders are more likely to be neglected from appropriate dementia care in time than the white counterparts. Among minorities group, Korean Americans (KAs) are the 4th largest and one of the most rapidly growing Asian subpopulations and have been characterized as under-resourced and underserved population of dementia care. This research is being done to understand how an education and navigation support program led by trained community health workers (CHWs) helps Korean American elders with probable dementia and the Korean American elders' caregivers. In a 2-arm randomized controlled trial (RCT) with 288 dyads, the investigators' aims are to (1) test the effect of a community-based intervention delivered by trained CHWs for undiagnosed KA elders with probable dementia and the KA elders' caregivers, (2) evaluate the effect of the PLAN on improving caregiver's dementia literacy, self-efficacy in dementia care and service use, social support, depression, and quality of life at 6 months in comparison to usual care, and (3) examine whether the effect of PLAN differs across age, sex, English proficiency and education caregiver subgroups. Exploratory Aim 1 is to test the effect of PLAN on Korean elders with probable dementia and caregiver development of a plan regarding dementia care at 6 months in comparison to usual care. The other two Exploratory Aims are to test the applicability of this study in another environment: Exploratory Aim 2: Using an equity-informed human-centered design framework, scale PLAN for implementation in ethnic daycare and Exploratory Aim 3: Pilot test the feasibility and acceptability of PLAN in ethnic adult daycare.

Aim 1 and Exploratory Aim test the following hypotheses: (1) Korean elders with probable dementia who receive the PLAN will have higher rates of linkage to medical service for dementia than those in the control group (Aim 1) and (2) Korean elders with probable dementia and the KA elders' caregivers who receive the PLAN will have higher rates of having a plan for dementia care than those in the control group (Exploratory Aim). Aim 2 tests the following hypothesis: Caregivers in the PLAN group will have higher dementia literacy, self-efficacy in dementia care and service use, social support, and quality of life, and lower depression than those in the control group.

ELIGIBILITY:
Patient Inclusion Criteria:

* Self-identified as first-generation KA
* Age 65 years or older
* CDR 1.0+
* Has a caregiver who lives in the same household or has at least weekly interactions
* Able to consent or has a proxy available for consent
* Written consent to participate in the study

Caregiver Inclusion Criteria:

* Age 18 years or older
* Able to read and speak Korean
* Lives in the same household with the elder or has at least weekly interactions
* Written consent to participate in the study and to allow the team to audit medical records for linkage to medical service for dementia

Patient Exclusion Criteria:

* Previous diagnosis of dementia
* All Axis I diagnoses other than depressive disorders (e.g., schizophrenia, bipolar disorder, or substance use disorder)
* Neurological disorders other than Alzheimer's disease that might affect cognition (e.g., stroke)
* Use of psychotropic drugs including antipsychotics,

Caregiver Exclusion Criteria:

* Plan to move from the area within 6 months
* Active treatment for a terminal illness or in hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants linked to medical service for dementia measured by medical record verification | 6 months
  Linkage to medical service for dementia is defined as the completion of a medical clinic visit by a Korean older adult with probable dementia.

SECONDARY OUTCOMES:
Caregiver's dementia literacy measured by dementia literacy test | 6 months
  Dementia literacy test is a 11-item instrument (true or false). Scoring of the dementia literacy instrument is in such a way that each correct response will be coded as 1 whereas incorrect response will be coded as 0. Total scores can range from 0 to 11 with higher scores indicating higher health literacy.
Self-efficacy in dementia care measured by dementia self-efficacy scale | 6 months
  Dementia self-efficacy scale is a 10-item instrument. Scoring of the dementia self-efficacy scale ranges from "not at all certain" coded as 1 to "very certain" coded as 10 for each item. Total scores will range from 10 to 100 with higher scores indicating higher self-efficacy.
Social support status as assessed by medical outcomes study scale | 6 months
  The 8-item scale of medical outcomes study scoring ranges from "none of the time" coded as 1 to "all of the time" coded as 5 for each item. Total scores will range from 8 to 40 with higher scores indicating higher social support.
Depression status as assessed by Patient Health Questionnaire-9 | 6 months
  Patient health questionnaire-9 is a 9-item instrument and scoring ranges from "not at all" coded as 0 to "nearly every day" coded as 3. Total scores will range from 0 to 27 with higher score indicating higher depression.
Quality of life (QoL) measured by QoL-dementia caregiver instrument | 6 months
  QoL-dementia caregiver is a 13-item instrument and scoring ranges from "poor" coded as 1 to "excellent" coded as 4 for each item. Total scores will range from 13 to 52 with higher scores indicating higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD, RN, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Korean Community Services of Metropolitan New York, Bayside, New York
  - Korean Community Service Center of Greater Washington, Annandale, Virginia

REFERENCES:
- [Derived] Min D, Yun JY, Parslow C, Jajodia A, Han HR. Online-Based Recruitment Methods for Community-Dwelling Older Adults: Scoping Review and Lessons Learned From the PLAN Trial. J Med Internet Res. 2025 Feb 25;27:e55082. doi: 10.2196/55082. PMID 39998873
- [Derived] Han HR, Perrin N, Kwon SC, Joo J, Yun JY, Min D, Lee HB. PLAN-Dementia literacy education and navigation for Korean elders with probable dementia and their caregivers: Rationale, methods, and design of a community-based, randomized, controlled, multi-site clinical trial. Contemp Clin Trials. 2025 Jan;148:107771. doi: 10.1016/j.cct.2024.107771. Epub 2024 Nov 30. PMID 39622468
- [Derived] Han HR, Yun JY, Min D, Razaz M. Health literacy demand and attitudes toward COVID-19 prevention measures among Korean American older adults and their caregivers. BMC Public Health. 2024 Oct 23;24(1):2941. doi: 10.1186/s12889-024-20427-7. PMID 39443891
- [Derived] Baumeister A, Aldin A, Chakraverty D, Hubner C, Adams A, Monsef I, Skoetz N, Kalbe E, Woopen C. Interventions for improving health literacy in migrants. Cochrane Database Syst Rev. 2023 Nov 14;11(11):CD013303. doi: 10.1002/14651858.CD013303.pub2. PMID 37963101
- [Derived] Han HR, Min D, Yun JY, Joo JH, Lee HB, Kwon S. The impact of anti-Asian racism on routine activities and mental health among Korean American older adults and their caregivers. Front Public Health. 2023 Feb 22;11:958657. doi: 10.3389/fpubh.2023.958657. eCollection 2023. PMID 36908462
- See also: Alzheimer's Association brochure about signs of dementia and dementia treatment, which is publicly available in Korean. — http://www.alz.org/asian/overview.asp?nL=KO&dL=KO